CLINICAL TRIAL: NCT01042769
Title: A Safety and Efficacy Study to Evaluate the Potential of Aleglitazar to Reduce Cardiovascular Risk in Coronary Heart Disease (CHD) Patients With a Recent Acute Coronary Syndrome (ACS) Event and Type 2 Diabetes Mellitus (T2D)
Brief Title: A Study With Aleglitazar in Patients With a Recent Acute Coronary Syndrome and Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC22140; 2009-012269-71
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar (Experimental)
  Interventions: Drug: Aleglitazar
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aleglitazar — aleglitazar 150 micrograms po daily
  Arms: Aleglitazar
Drug: Placebo — placebo control po daily
  Arms: Placebo

SUMMARY:
This double-blind, parallel, two-arm study will evaluate the potential to reduce cardiovascular risk, the tolerability and long-term safety profile of aleglitazar compared to placebo on top of standard care in patients with recent acute coronary syndrome (ACS) and type 2 diabetes mellitus. Patients will be randomized to receive either aleglitazar or placebo once daily as oral doses. The study will last until at least 950 events occur, but time on study treatment will be for at least 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Type 2 diabetes mellitus
* Hospitalization for ACS event and randomization between hospital discharge and 8 weeks after the ACS index event (day of hospitalization)

Exclusion Criteria:

* Estimated glomerular filtration rate <45 mL/min/1.73m2
* Concomitant treatment with a thiazolidinedione and/or fibrate
* Triglycerides >400 mg/dL
* Anaemia
* Symptomatic congestive heart failure classified as New York Heart Association (NYHA) class II-IV (France and Germany: Symptomatic congestive heart failure classified as NYHA class I-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7226 (Actual)
Dates: Start 2010-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Effect on cardiovascular death, non-fatal myocardial infarction and non-fatal stroke | Throughout study, approximately 4.5 years

SECONDARY OUTCOMES:
Effects on other cardiovascular endpoints | Throughout study, approximately 4.5 years
Glycemic control, lipoprotein profile, blood pressure, biomarkers of cardiovascular risk | Throughout study, months 1, 3, 6, 9, 12 and then every 6 months thereafter
Tolerability and long-term safety profile | Throughout study, approximately 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (618):
- United States (184):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Banning, California
  - Carmichael, California
  - Fresno, California
  - Fullerton, California
  - Glendale, California
  - Hawaiian Gardens, California
  - Inglewood, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Northridge, California
  - Orange, California
  - Pomona, California
  - Redondo Beach, California
  - Salinas, California
  - San Diego, California
  - San Francisco, California
  - Santa Ana, California
  - Sylmar, California
  - Thousand Oaks, California
  - Torrance, California
  - Ventura, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Hartford, Connecticut
  - Stamford, Connecticut
  - Seaford, Delaware
  - Aventura, Florida
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Coral Springs, Florida
  - Doral, Florida
  - Edgewater, Florida
  - Elizabeth, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville Beach, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Miramar, Florida
  - Naples, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Panama City, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Trinity, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Gurnee, Illinois
  - Elkhart, Indiana
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Ames, Iowa
  - Council Bluffs, Iowa
  - Davenport, Iowa
  - Des Moines, Iowa
  - Elizabethtown, Kentucky
  - Owensboro, Kentucky
  - Alexandria, Louisiana
  - Convington, Louisiana
  - Hammond, Louisiana
  - Houma, Louisiana
  - Lafayette, Louisiana
  - Laplace, Louisiana
  - Metarie, Louisiana
  - New Orleans, Louisiana
  - Opelousas, Louisiana
  - Shreveport, Louisiana
  - Slidell, Louisiana
  - Zachary, Louisiana
  - Bangor, Maine
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Columbia, Maryland
  - Oxon Hill, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Hyannis, Massachusetts
  - Worcester, Massachusetts
  - Alpena, Michigan
  - Ann Arbor, Michigan
  - Bay City, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Petoskey, Michigan
  - Royal Oak, Michigan
  - Saginaw, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Jackson, Mississippi
  - Picayune, Mississippi
  - Chesterfield, Missouri
  - Washington, Missouri
  - Great Falls, Montana
  - Freemont, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Bridgewater, New Jersey
  - Mine Hill, New Jersey
  - Newark, New Jersey
  - Somerset, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Suffern, New York
  - Syracuse, New York
  - The Bronx, New York
  - Troy, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Rocky Mount, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Kettering, Ohio
  - Marion, Ohio
  - Middleburg Heights, Ohio
  - Springfield, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Chambersburg, Pennsylvania
  - Danville, Pennsylvania
  - Harrisburg, Pennsylvania
  - Natrona Heights, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottstown, Pennsylvania
  - Upper Darby, Pennsylvania
  - Pawtucket, Rhode Island
  - Providence, Rhode Island
  - Greer, South Carolina
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Lexington, Tennessee
  - Nashville, Tennessee
  - Tullahoma, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Bellaire, Texas
  - Dallas, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Kerrville, Texas
  - Kingwood, Texas
  - Lubbock, Texas
  - Odessa, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Victoria, Texas
  - Layton, Utah
  - Murray, Utah
  - Danville, Virginia
  - Roanoke, Virginia
  - Huntington, West Virginia
  - Beloit, Wisconsin
  - Burlington, Wisconsin
  - Green Bay, Wisconsin
  - La Crosse, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (16):
  - Buenos Aires
  - Caba
  - Capital Federal
  - Ciudad Autonoma Bs As
  - Coronel Suárez
  - Corrientes
  - Córdoba
  - Haedo
  - Mendoza
  - Morón
  - Rosario
  - Salta
  - San Miguel de Tucumán
  - Santa Fe
  - Santiago del Estero
  - Zárate
- Australia (22):
  - Garran, Australian Capital Territory
  - Bankstown, New South Wales
  - Concord, New South Wales
  - Darlinghurst, New South Wales
  - Liverpool BC, New South Wales
  - New Lambton, New South Wales
  - Penrith, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Wollongong, New South Wales
  - Douglas, Queensland
  - Milton, Queensland
  - Redcliffe, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Elizabeth Vale, South Australia
  - Woodville, South Australia
  - Ballarat, Victoria
  - Geelong, Victoria
  - Richmond, Victoria
  - Shepparton, Victoria
- Brazil (20):
  - Fortaleza, Ceará
  - Cariacica, Espírito Santo
  - Salvador, Estado de Bahia
  - Brasília, Federal District
  - Goiânia, Goiás
  - Campo Grande, Mato Grosso do Sul
  - Belo Horizonte, Minas Gerais
  - Uberlândia, Minas Gerais
  - Campina Grande do Sul, Paraná
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Natal, Rio Grande do Norte
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Sao Jose Do Rio Preto, Santa Catarina
  - São José, Santa Catarina
  - Campinas, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
- Canada (45):
  - Edmonton, Alberta
  - Red Deer, Alberta
  - New Westminster, British Columbia
  - Surrey, British Columbia
  - Bathurst, New Brunswick
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Bridgewater, Nova Scotia
  - Halifax, Nova Scotia
  - Brampton, Ontario
  - Burlington, Ontario
  - Cambridge, Ontario
  - Fort Eire, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Smiths Falls, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Charlottetown, Prince Edward Island
  - Chicoutimi, Quebec
  - Gatineau, Quebec
  - Granby, Quebec
  - Laval, Quebec
  - Lévis, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Jérôme, Quebec
  - Saint-Lambert, Quebec
  - Saint-Laurent, Quebec
  - Saint-Léonard, Quebec
  - Sherbrooke, Quebec
  - Ste. Foy, Quebec
  - Terrebonne, Quebec
  - Trois-Rivières, Quebec
  - Val DOr, Quebec
  - Vaudreuil-Dorion, Quebec
- China (19):
  - Baotou
  - Beijing
  - Beijng
  - Changsha
  - Chengdu
  - Dalian
  - Daqing
  - Guangzhou
  - Hangzhou
  - Jinan
  - Nanjing
  - Nanning
  - Qingdao
  - Shanghai
  - Shenyang
  - Shijiazhuang
  - Tianjin
  - Wuhan
  - Xi'an
- Czechia (10):
  - Brno
  - Hradec Králové
  - Jindřichův Hradec
  - Kladno
  - Olomouc
  - Prague
  - Tábor
  - Teplice
  - Trutnov
  - Znojmo
- Denmark (6):
  - Aalborg
  - Copenhagen
  - Fredericia
  - Herning
  - Odense
  - Slagelse
- France (16):
  - Albi
  - Besançon
  - Bron
  - Cambrai
  - Créteil
  - Dijon
  - Lagny-sur-Marne
  - Le Coudray
  - Le Plessis-Robinson
  - Marseille
  - Montfermeil
  - Montpellier
  - Paris
  - Pessac
  - Saint-Herblain
  - Valenciennes
- Germany (36):
  - Bad Krozingen
  - Bad Nauheim
  - Bad Oeynhausen
  - Bad Rothenfelde
  - Berlin
  - Bernried
  - Bochum
  - Bonn
  - Brandenburg
  - Burg
  - Cologne
  - Dortmund
  - Düsseldorf
  - Essen
  - Frankfurt
  - Fulda
  - Fürth
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Homburg/Saar
  - Kiel
  - Lahr
  - Langen
  - Mainz
  - Mannheim
  - Mönchengladbach
  - München
  - Münster
  - Nienburg
  - Pirna
  - Regensburg
  - Rotenburg (Wümme)
  - Rüdersdorf
  - Wuppertal
- Toulouse, Grenada
- Hungary (12):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Gyula
  - Kaposvár
  - Kecskemét
  - Miskolc
  - Pécs
  - Székeshehérvár
  - Szolnok
  - Szombathely
  - Zalaegerszeg
- India (24):
  - Kochi, Kerala
  - Pune, Maharashtra
  - Ahmedabad
  - Bangalore
  - Banglore
  - Belagavi
  - Chennai
  - Gūrgaon
  - Hyderabad
  - Indore
  - Jaipur
  - Kochi
  - Kolkata
  - Lucknow
  - Madurai
  - Mangalore
  - Mumbai
  - Mysore
  - Nagpur
  - New Delhi
  - Palakkad
  - Pune
  - Secunderabad
  - Trivandeum
- Ireland (4):
  - Ballinasloe
  - Dublin
  - Galway
  - Tallaght Dublin
- Italy (15):
  - Napoli, Campania
  - Pozzuoli, Campania
  - Bentivoglio, Emilia-Romagna
  - Ferrara, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Bergamo, Lombardy
  - Legnano, Lombardy
  - Mantova, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
  - Perugia, Umbria
  - Cittadella, Veneto
  - Rovigo, Veneto
- Malaysia (7):
  - Sarawak, Sarawak
  - George Town
  - Kelantan
  - Kota Bharu
  - Kuala Lumpur
  - Kuantan
  - Serdang
- Mexico (21):
  - Acapulco
  - Aguascalientes
  - Chihuahua City
  - Ciudad Juárez
  - Cuernavaca
  - Culiacán
  - Durango
  - Guadalajara
  - Mexico City
  - Monterrey
  - Pachuca
  - Puebla City
  - Puerto Vallarta
  - Querétaro
  - San Luis Potosi S.l.p.
  - Tampico
  - Tijuana
  - Tlalnepantla
  - Veracruz
  - Xalapa
  - Zapopan
- Netherlands (13):
  - AC Amsterdam
  - Amstelveen
  - Amsterdam
  - Hoorn
  - Leiden
  - Maastricht
  - Nieuwegein
  - Nijmegen
  - Purmerend
  - Tilburg
  - Weert
  - Zaandam
  - Zwolle
- New Zealand (7):
  - Auckland
  - Christchurch
  - Hamiton
  - Lower Hutt
  - Nelson
  - Palmerston North
  - Tauranga
- Poland (38):
  - Bêdzin
  - Bialystok
  - Bielsko-Biala
  - Bydgoszcz
  - Bytom
  - Gdansk
  - Gdynia
  - Gorlice
  - Grodzisk Mazowiecki
  - Katowice
  - Kędzierzyn-Koźle
  - Kielce
  - Krakow
  - Kutno
  - Libiąż
  - Lodz
  - Lublin
  - Nowa Sól
  - Nysa
  - Olesnica, Spalice
  - Olsztyn
  - Oława
  - Poznan
  - Puławy
  - Radom
  - Rzeszów
  - Swidnica
  - Tarnów
  - Torun
  - Ustroń
  - Ustroñ
  - Warsaw
  - Wola
  - Wroclaw
  - Zamość
  - Zgorzelec
  - Żarów
  - £ódx
- Romania (10):
  - Brasov
  - Bucharest
  - Buzău
  - Cluj-Napoca
  - Craiova
  - Galati
  - Oradea
  - Ploieşti
  - Târgu Mureş
  - Timișoara
- Russia (2):
  - Moscow
  - Saint Petersburg
- South Korea (13):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Jeollabuk-do
  - Kyonggi-do
  - Seoul
  - Suwon
  - Uijongbu
  - Ulsan
  - Wŏnju
- Spain (28):
  - Vitoria-Gasteiz, Alava
  - Alicante, Alicante
  - Torrevieja, Alicante
  - Almería, Almeria
  - Barcelona, Barcelona
  - Granollers, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Sabadell, Barcelona
  - Terrassa, Barcelona
  - Jerez de la Frontera, Cadiz
  - Figueres, Girona
  - Guadalajara, Guadalajara
  - A Coruña, La Coruña
  - Ferrol, La Coruña
  - Santiago de Compostela, La Coruña
  - Lugo, Lugo
  - Alcorcón, Madrid
  - Madrid, Madrid
  - San Sebastián de los Reyes, Madrid
  - Málaga, Malaga
  - Murcia, Murcia
  - Oviedo, Principality of Asturias
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Reus, Tarragona
  - Tarragona, Tarragona
  - Valencia, Valencia
  - Bilbao, Vizcaya
- Sweden (11):
  - Danderyd Stockholm
  - Gothenburg
  - Halmstad
  - Kalmar
  - Karlstad
  - Kristianstad
  - Malmo
  - Östersund
  - Skellefteå
  - Skövde
  - Stockholm
- Thailand (10):
  - Amphur Mae-Rim
  - Amphur Muang
  - Bangkok
  - Changwat Sara Buri
  - Chiang Mai
  - Chon Buri
  - Khon Kaen
  - Khonkaen
  - Klong Luang
  - Phitsanulok
- United Kingdom (28):
  - Abano Terme
  - Antrim
  - Ayr
  - Basildon
  - Bath
  - Belfast
  - Brighton
  - Cambridge
  - Craigavon
  - Derby
  - Glasgow
  - Harrow
  - Inverness
  - Isle of Wight
  - Isleworth
  - Leeds
  - London
  - Manchester
  - Middlesex
  - Newcastle upon Tyne
  - Northampton
  - Paddington
  - Plymouth
  - Poole
  - Romford
  - Stoker on Trent
  - West Bromwich
  - Wrexham

REFERENCES:
- [Derived] Schrieks IC, Nozza A, Stahli BE, Buse JB, Henry RR, Malmberg K, Neal B, Nicholls SJ, Ryden L, Mellbin L, Svensson A, Wedel H, Weichert A, Lincoff AM, Tardif JC, Grobbee DE, Schwartz GG. Adiponectin, Free Fatty Acids, and Cardiovascular Outcomes in Patients With Type 2 Diabetes and Acute Coronary Syndrome. Diabetes Care. 2018 Aug;41(8):1792-1800. doi: 10.2337/dc18-0158. Epub 2018 Jun 14. PMID 29903845
- [Derived] Lincoff AM, Tardif JC, Schwartz GG, Nicholls SJ, Ryden L, Neal B, Malmberg K, Wedel H, Buse JB, Henry RR, Weichert A, Cannata R, Svensson A, Volz D, Grobbee DE; AleCardio Investigators. Effect of aleglitazar on cardiovascular outcomes after acute coronary syndrome in patients with type 2 diabetes mellitus: the AleCardio randomized clinical trial. JAMA. 2014 Apr 16;311(15):1515-25. doi: 10.1001/jama.2014.3321. PMID 24682069
- [Derived] Lincoff AM, Tardif JC, Neal B, Nicholls SJ, Ryden L, Schwartz GG, Malmberg K, Buse JB, Henry RR, Wedel H, Weichert A, Cannata R, Grobbee DE. Evaluation of the dual peroxisome proliferator-activated receptor alpha/gamma agonist aleglitazar to reduce cardiovascular events in patients with acute coronary syndrome and type 2 diabetes mellitus: rationale and design of the AleCardio trial. Am Heart J. 2013 Sep;166(3):429-34. doi: 10.1016/j.ahj.2013.05.013. Epub 2013 Jul 26. PMID 24016490